CLINICAL TRIAL: NCT07245602
Title: Biomechanical Study on the Improvement of Lower Limb Motor Function in the Elderly Through Collaborative Functional Electrical Stimulation
Brief Title: A Biomechanical Study of Collaborative FES on Lower Limb Motor Function in the Elderly
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chen Xuan (Other)
Responsible Party: Sponsor-Investigator, Chen Xuan, graduate student, Southern Medical University, China
Organization: Southern Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202551
Record Dates: First submitted 2025-09-25; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Muscle Fatigue (C23.888.592.612.612); Muscle Weakness or Atrophy
MeSH Terms: conditions — Muscle Weakness; Atrophy

STUDY DESIGN:
Who Masked: Participant
Masking Description: This study will employ a single-blind (assessor-blinded) design.
  Participants and Therapists: Due to the distinct nature of the two electrical stimulation interventions, blinding of participants and the therapists administering the treatments is not feasible. However, to minimize expectation bias, all participants will be informed that they will be randomized to one of two "effective" types of electrical stimulation therapy, without disclosing the specific differences between them.
  Outcome Assessors: All primary and secondary outcome measures will be collected by an independent assessor who is blinded to the group allocation of the participants. This assessor will not be involved in the intervention process and will be strictly instructed to refrain from discussing any treatment-related information with the participants or therapists throughout the study.
  Data Analysts: During the data analysis phase, the two groups will be coded as "Group A" and "Group B". The data analyst will per
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm: Conventional Functional Electrical Stimulation (Placebo Comparator): Participants will receive functional electrical stimulation (FES) administered in a conventional, non-synergy-based mode. This arm serves as an active comparator.
  Interventions: Device: Traditional functional electrical stimulation
- Experimental Arm: Muscle Synergy-Based Functional Electrical Stimulation (Experimental): Participants will receive a novel functional electrical stimulation (FES) intervention guided by a real-time, muscle synergy-based algorithm.
  Interventions: Device: Collaborative Functional Electrical Stimulation

INTERVENTIONS:
Device: Collaborative Functional Electrical Stimulation — Functional electrical stimulation based on muscle synergy
  Arms: Experimental Arm: Muscle Synergy-Based Functional Electrical Stimulation
Device: Traditional functional electrical stimulation — Traditional functional electrical stimulation
  Arms: Control Arm: Conventional Functional Electrical Stimulation

SUMMARY:
This study will first conduct a precise assessment of the differences in muscle coordination among the elderly through muscle synergy analysis; then, based on this, it will extract abnormal synergy patterns and muscle activation patterns, and reconstruct the intervention's synergy modules to fit the intervention electrostimulation curve; finally, electrical stimulation interventions will be carried out on different elderly individuals under two conditions: sitting and walking, to evaluate the intervention effects and analyze the biomechanical mechanisms of its effectiveness.

DETAILED DESCRIPTION:
The research subjects of this project mainly focus on young people, middle-aged individuals, and elderly individuals who are able to move independently. The investigator's goal is to explore the kinematic and dynamic characteristics of different populations. The main research activities include recruiting young volunteers, middle-aged volunteers, and elderly volunteers who can move independently. Through motion capture, the kinematic data and surface electromyography (sEMG) signal confidence intervals of young and middle-aged subjects are analyzed, and then the kinematic data and sEMG data of independently mobile elderly individuals are examined. The investigator aims to identify multiple muscles that show significant differences compared to normal individuals, and then assess the effectiveness of functional electrical stimulation based on coordinated movement. Additionally, using in vivo motion technology, the investigator will establish a human biomechanics database to analyze the biomechanical characteristics of different populations under various movement conditions.

ELIGIBILITY:
Inclusion Criteria:

* Must be aged between 65 and 75 years, inclusive.
* Must be community-dwelling.
* Must be able to ambulate independently, with or without the use of an assistive device (e.g., a cane or walker).
* Must be capable of understanding and following study-related instructions and procedures.
* Must provide voluntary written informed consent to participate in the study.

Exclusion Criteria:

* Diagnosis of a significant neurological disorder, including but not limited to stroke, Parkinson's disease, or multiple sclerosis.
* Presence of a severe musculoskeletal condition that would interfere with movement tasks, such as severe osteoarthritis or osteoporosis.
* History of lower limb joint replacement surgery within the last 6 months.
* Cognitive impairment, as indicated by a Mini-Mental State Examination (MMSE) score of less than 24.
* Presence of any implanted electronic medical device, such as a cardiac pacemaker or defibrillator.
* Any skin disease, open wound, infection, or malignancy at the intended sites of electrical stimulation.
* Diagnosis of a severe and/or uncontrolled cardiovascular condition (e.g., unstable angina, recent myocardial infarction).
* Inability to stand independently without support for at least 3 minutes.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Muscle electrical signals | On the first day of the study, muscle electrical signals were tested using electromyography equipment. After one month of intervention, these indicators were measured again, followed by a one-year follow-up with the participants until the study ended.
  Electromyographic signals were collected from 16 muscles of the trunk and ipsilateral leg using a wireless EMG system (Mini Wave Infinity by Cometa, Italy) at a frequency of 2000 Hz, with an interelectrode distance of 20 mm.
Important indicators kinematic data | On the first day of the study, kinematic data, including joint angles and stride length, were collected using the Qualisys gait analysis system. After one month of intervention, these measurements were taken again
  Attach Mark points to the subjects and capture kinematic data through an infrared camera.The movement of the foot and lower limb joints was captured using eight optical infrared cameras (also sampled at 100 Hz; Miqus M1, Qualisys, Sweden) and one camera lens (Miqus Video, Qualisys, Sweden), calculating the positions of 56 optical markers.

SECONDARY OUTCOMES:
Secondary indicators | On the first day of the study, foot pressure was measured using a plantar pressure testing mat, followed by a one-month intervention, after which the same indicators were measured again. Subsequently, the subjects were followed up for one year
  Plantar pressure, distribution of plantar pressure on the left and right feet at rest, and distribution of pressure intensity on the left and right feet while walking

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Chen, Study Chair — Southern Medical University

IPD SHARING:
Plan to Share IPD: No